CLINICAL TRIAL: NCT06449508
Title: Role of Probiotics Administered as an Adjuvant Therapy in Pathological Neonatal Unconjugated Hyperbilirubinemia
Brief Title: The Effectiveness of Probiotics in Neonatal Jaundice
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Samah Safwat, Principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Probiotics in jaundice
Record Dates: First submitted 2024-06-01; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Jaundice, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal | interventions — Lacteol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): no intervention
- probiotics (Active Comparator): will receive 5 drops of probiotic supplement containing Bacillus clausil spores (Enterogermania amp 2 billion/5 mL) once daily plus phototherapy till discharge.
  Interventions: Drug: Probiotic Formula

INTERVENTIONS:
Drug: Probiotic Formula — drops of probiotic supplement containing bacillus clausil spores (Enterogermania Amp 2 Billion/5Ml )
  Other Names: lactobacillus
  Arms: probiotics

SUMMARY:
Hyperbilirubinemia is a prevalent problem in babies that necessitates medical attention. Probiotic administration as adjuvant therapy may have a positive impact on the pathological neonatal unconjugated hyperbilirubinemia.

DETAILED DESCRIPTION:
Neonatal jaundice is a common health care issue that affects approximately 9% of newborns after birth. The percent of neonates who acquire jaundice in the first week of their birth is about 60%. while the percent of breasted neonates who develop jaundice during the first month of their birth is about 10%.

Phototherapy is the standard therapy for neonates who develop pathological jaundice, as it can alter bilirubin structure and increase its excretion.

Probiotics can also be used for the treatment of jaundice. The efficacy of probiotics depends on their ability to pass across the GIT and cause colonization in the intestinal lumen. Hence, it leads to a decrease in the bacterial growth in the small bowel, a reduction in the function of the gastrointestinal barrier, and a regulation of the immune system of the host.

ELIGIBILITY:
Inclusion Criteria:

* Neonate suffered from pathological unconjugated hyper-bilirubinemia with Total serum bilirubin (TSB) between 5-15mg/dl and need phototherapy.

Exclusion Criteria:

* neonates who have kernicterus.
* neonates who have ventilation problem.
* neonates who have heart failure.
* -neonates who have asphyxia.
* neonates who have history of Rh incompatibility

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
the change in the measured total bilirubin, direct bilirubin, and Indirect Bilirubin. | up to 4 weeks

SECONDARY OUTCOMES:
The change in serum concentration of the Human Tumor Necrosis Factor Alpha (TNFa) | up to 4weeks

IPD SHARING:
Plan to Share IPD: No